CLINICAL TRIAL: NCT04479774
Title: Effects of Compelled Body Weight Shift Technique for Rehabilitation of Individuals With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwest Institute of Health Sciences, Pakistan (Other)
Responsible Party: Principal Investigator, Usman Farooq, Dr.Usman Farooq PT, Northwest Institute of Health Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NWIHS-0001/IRB/01
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Chronic Stroke
Keywords: compelled body shift technique; stroke; tinetti performance oriented mobility assessment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Participants random allocation into control and experimental groups
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Group A) (Experimental): Subjects were randomly assigned and informed consent was obtained, the subjects were educated about treatment and on the basis of functional ambulation scale 3,4 and 5 subjects were included, along with this the subjects of age group between 40-60 having ability to understand and follow instructions were included in study.
  Results were obtained by using gait parameters including walk speed, cadence, step rate, stride length The tinetti POMA scale was utilized to record changes post treatment in gait , the weight bearing was recorded using Camry ZT-160 analog weight scale At the end of every week results were obtained.
  Interventions: Other: Compelled Body Weight Shift Technique
- Control group: (Group B) (Other): Subjects were randomly assigned and informed consent was obtained, the subjects were educated about treatment and on the basis of functional ambulation scale 3,4 and 5 subjects were included, along with this the subjects of age group between 40-60 having ability to understand and follow instructions were included in study.
  Results were obtained by using gait parameters including walk speed, cadence, step rate, stride length The tinetti POMA scale was utilized to record changes post treatment in gait , the weight bearing was recorded using Camry ZT-160 analog weight scale At the end of every week results were obtained.
  Interventions: Other: Compelled Body Weight Shift Technique without insole

INTERVENTIONS:
Other: Compelled Body Weight Shift Technique — Routine Physical Therapy with 0.6 cm thickness insole inserted in shoe of unaffected side and following exercises were performed by patients
  * Muscle re-education
  * Sit to stand exercise , 4 to 10 repetitions
  * Supported heel raise to 10 repetitions with 3 sets
  * Supported squat exercise tibialis anterior and quads muscles to 10 repetitions with 3 sets
  * Gait training
  * Forward walk in parallel bars with number of 10 rounds.
  * Task oriented training balance training
  * A. Stepping exercise on 15 cm height step and number of repetitions 10.
  * B. Tandem standing for 10 seconds.
  * C. Reaching exercise in which patient performed reaching for object in therapists hand and the number of repetitions was 10.
  Arms: Experimental Group (Group A)
Other: Compelled Body Weight Shift Technique without insole — Routine Physical Therapy without 0.6 cm thickness insole inserted in shoe of unaffected side and following exercises were performed by patients
  * Muscle re-education
  * Sit to stand exercise , 4 to 10 repetitions
  * Supported heel raise to 10 repetitions with 3 sets
  * Supported squat exercise tibialis anterior and quads muscles to 10 repetitions with 3 sets
  * Gait training
  * Forward walk in parallel bars with number of 10 rounds.
  * Task oriented training balance training
  * A. Stepping exercise on 15 cm height step and number of repetitions 10.
  * B. Tandem standing for 10 seconds.
  * C. Reaching exercise in which patient performed reaching for object in therapists hand and the number of repetitions was 10.
  Arms: Control group: (Group B)

SUMMARY:
Stroke is one of the major cause of lifelong disability if not treated on time, the investigator's technique knows as Compelled Body Weight Shift Technique (CBWS) was utilized and administered to chronic stroke population and results were figured out using gait parameters and Tinetti POMA scale.

DETAILED DESCRIPTION:
Total 28 sample size out of which 27 were divided into control and experimental group. Inclusion criteria was Unilateral chronic stroke with asymmetrical stance, Patients with score of 3,4 and 5 will be included according to FAS (Functional Ambulation Scale), Ability to understand and follow instructions, Both male and female, Any type of stroke, and Age 40-60. Written and informed consent was obtained from participants of study. Six weeks of exercise training was combined with compelled body weight shift technique via shoe lift of 0.6 cm thickness for experimental group and for control group training was performed without shoe lift.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral chronic stroke with asymmetrical stance
* Patients with score of 3,4 and 5 were included according to functional ambulation scale(59)
* Ability to understand and follow instruction
* Both male and female.
* Any type of stroke.
* Age 40-60.

Exclusion Criteria:

* • Serious or unstable medical, condition of patient.

  * History of other neurological diseases (i.e. Parkinson's disease, multiple sclerosis),
  * Contractures or any deformity.
  * Leg Length Discrepancy

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2020-07-12 (Actual); Primary Completion 2020-08-29 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Tinetti Performance Oriented Mobility Assessment | upto 6 weeks
  Tinetti Performance Oriented Mobility Assessment The Tinetti, evaluation instrument is, an effectively managed, task-arranged test that, quantifies gait and balance activities of patients. A three-point, ordinal scale, extending from 0-2. "0" demonstrates the most elevated level of debilitation and "2" the people's freedom.
  1. Total Balance Score = 16
  2. Total Gait Score = 12
  3. Maximum total test Score = 28 [Time Frame: upto 6 weeks]

SECONDARY OUTCOMES:
A 10meter walk test | upto 6 weeks
  A 10meter walk test A ten meter distance employed, to determine functional mobility and gait speed, the ten meter walk test was performed by patient at self-selected walking pace and fast walking pace
Camry 160 Analog Weight Scale | upto 6 weeks
  Camry 160 Analog Weight Scale to check the weight in kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- Usman Farooq, Mspt, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code